CLINICAL TRIAL: NCT01734343
Title: Posterior Capsule Opacification Development and Frequency of Nd:YAG Treatment of Two Microincision IOLs: Hoya iMics Y-60H vs. PhysIOL microAY
Brief Title: Posterior Capsule Opacification Development With Two Different Intraocular Lenses
Acronym: MIPHY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Rupert Menapace, Ao.Univ.-Prof. Dr.med.univ., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: EK Nr:847/2010
Record Dates: First submitted 2012-11-22; First posted 2012-11-27 (Estimated); Last update posted 2012-11-27 (Estimated); Status verified 2012-11

CONDITIONS: Posterior Capsule Opacification; Cataract
Keywords: posterior capsule opacification; PCO; after cataract; intraocular lens
MeSH Terms: conditions — Cataract; Capsule Opacification

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- HOYA iMics Y-60H (Other): eyes with implanted intraocular lens HOYA iMics Y-60H
  Interventions: Device: HOYA iMics Y-60H
- PhysIOL microAY (Other): eyes with implanted intraocular lens PhysIOL microAY
  Interventions: Device: PhysIOL microAY

INTERVENTIONS:
Device: HOYA iMics Y-60H — same-day bilateral cataract surgery with implantation of intraocular lens HOYA iMics Y-60H in one eye
  Arms: HOYA iMics Y-60H
Device: PhysIOL microAY — same-day bilateral cataract surgery with implantation of intraocular lens PhysIOL microAY in one eye
  Arms: PhysIOL microAY

SUMMARY:
Age-related cataract is the main cause of impaired vision in the elderly population worldwide.

The only treatment that can restore functional visual ability is cataract surgery where the opacified crystalline lens is removed by phacoemulsification and an artificial intraocular lens is implanted into the remaining capsular bag. Cataract operations are generally very successful, with a low risk of serious complications.

The most common reason for impaired vision after uneventful cataract surgery in otherwise healthy eyes is the development of posterior capsule opacification (PCO). PCO is a physiological change (thickening, opacification and clouding) of the capsular bag expected after cataract surgery, because the lens epithelial cells (LECs) undergo hyperplasia and cellular migration. PCO is treated with Nd:YAG capsulotomy, a quick outpatient procedure that uses a laser to open a central hole in the posterior capsular bag.

Modifications in IOL design and material lead to a decrease in the incidence of PCO.

During the past two decades, refinements in surgical technique were made resulting in today's small incision phacoemulsification surgery. Nowadays a multitude of microincision IOLs are available, many of them similar but of course with some differences in regard to the chemical composition of the acrylic material and the IOL design.

The purpose of this study is to compare the development of posterior capsule opacification (PCO) and the frequency of treatment between two different microincision IOLs over a period of 3 years.

ELIGIBILITY:
Inclusion Criteria:

* bilateral age-related cataract
* good overall physical constitution

Exclusion Criteria:

* previous intraocular surgery or ocular trauma
* intraocular complication like posterior capsular tear
* glaucoma
* uveitis
* corneal diseases, diabetic retinopathy and any other severe retinal pathology that would make a postoperative visual acuity of 20/40 (decimal equivalent = 0.5) or better unlikely

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2009-01; Primary Completion 2012-05 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
posterior capsular opacification (PCO) | 3 years
  subjective and objective PCO scoring

SECONDARY OUTCOMES:
best corrected visual acuity (BCVA) | 3 years
Nd:YAG rate | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Rupert Menapace, Prof. Dr., Principal Investigator — Medical University of Vienna
Locations (1):
- Department of Ophthalmology and Optometry of the Medical University Vienna, Vienna, Vienna, Austria